CLINICAL TRIAL: NCT03024801
Title: Effectiveness of Autologous Platelet-rich Plasma on Knee Cartilage Injury: a Randomized, Controlled, Open-label Clinical Trial
Brief Title: Effectiveness of Autologous Platelet-rich Plasma on Knee Cartilage Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanyi Guo, Chief Physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLAGH_003
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Cartilage Injury
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- autologous platelet-rich plasma group (Experimental): The patients with knee cartilage injury were randomized to the intra-articular injection of autologous platelet-rich plasma group.
  Interventions: Drug: autologous platelet-rich plasma
- normal saline group (Experimental): The patients with knee cartilage injury were randomized to the normal saline group.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: autologous platelet-rich plasma — The patients with knee cartilage injury were randomized to the intra-articular injection of autologous platelet-rich plasma group.
  Arms: autologous platelet-rich plasma group
Drug: normal saline — The patients with knee cartilage injury were randomized to the normal saline group.
  Arms: normal saline group

SUMMARY:
To analyze the effectiveness of intra-articular injection of autologous PRP on knee cartilage repair and evaluating functional recovery of the knee joint in knee cartilage injury patients.

DETAILED DESCRIPTION:
Recent studies have shown that platelets, which contain a large number of cytokines and growth factors, can be beneficial in inflammatory response and postoperative bleeding, infection, bone formation, injury, muscle strain, and soft tissue healing. Platelets release a plethora of biologically active proteins to aggregate macrophages, mesenchymal stem cells (MSCs) and osteoblasts, thereby promoting degradation and clearing necrotic tissue, thus further activating wound healing. In fact, platelet-rich plasma (PRP) is now used clinically to promote cartilage repair.

By retrieving the Web of Science, a study by Havva et al. reported the clinical use of autologous PRP in 82 patients with advanced knee osteoarthritis with good outcomes. However, the clinical applications of this treatment have not been adequately investigated in randomized controlled trials. Given this, additional studies on the exact efficacy of this treatment are indispensible.

Three similar trial protocols to the current trial include 'Treatment of Osteoarthritis by Intra-articular Injection of Bone Marrow Mesenchymal Stem Cells With Platelet Rich Plasma (NCT02365142)', 'PRP vs HA Intra-articular Knee Injections for Cartilage Defects (NCT02012530)', and 'Mesenchymal Stem Cells Enhanced With PRP Versus PRP In OA Knee (MSCPRPOAK) (NCT01985633)'. In these trial protocols, knee injury extent and treatment success were assessed by Osteoarthritis Score, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Visual Analog Scale (VAS) score as outcome measures. However, there are several differences in the inclusion criteria and randomization of these trials in comparison with the current trial protocol.

Since autologous PRP predominantly functions to relieve pain and inhibit inflammatory responses, clinical injection of autologous PRP for cartilage injury can stimulate chondrocyte growth and matrix metabolism. Existing evidence has shown that autologous PRP can increase type II collagen production and reduce apoptosis in chondrocytes when combined with autologous bone marrow-MSCs. Furthermore, PRP can improve cartilage degeneration and inhibit the development of osteoarthritis (OA) when combined with hydrogel microspheres. Accordingly, the clinical use of autologous PRP can alleviate the symptoms of OA, promote recovery of motor function, and ultimately improve patient quality of life.

To date, the clinical use of low-dose autologous PRP has been reported to alleviate pain at the injury site in the treatment of articular cartilage injury, and achieve cartilage repair and proliferation by releasing growth factors that promote extracellular matrix synthesis and vascular reconstruction. However, the clinical applications of autologous PRP have not been systemically reported in randomized controlled clinical trials, leading to a lack of objective evidence on its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Knee cartilage injury
* Having normal and stable joint motion but no deformity
* Focal cartilage defects confirmed by magnetic resonance imaging (MRI), Outerbridge classification III/IV with a defect size < 10 cm2 graded as Outerbridge II at maximum
* Focal articular cartilage injury in the knee
* 14-55 years of age
* Provision of signed informed consent to participate in the trial

Exclusion Criteria:

* Poor general condition
* Blood diseases
* Use of local hormone treatment within 3 months before the trial
* Bleeding tendency
* Drug addiction, including anesthetic, alcohol and poison
* Inflammatory arthropathy, including specific and non-specific arthritis and severe osteoarthritis
* Contagious viral infection
* Metabolic diseases, such as gout and rheumatism
* Pregnant or lactating, or planning to become pregnant within 1 year after the initial registration
* Unable to cooperate with rehabilitation therapy because of psychological/mental disorders

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lysholm score | at 3 months after final injection
  To assess functional recovery of the knee joint. Lysholm score ranges from 0-100 with higher scores indicating better knee joint function. A score <70 indicates damage to the knee joint function.

SECONDARY OUTCOMES:
2000 IKDC Subjective Knee Evaluation Form score | at 3 months after final injection
  To used for assessing functional recovery of the knee joint. Higher scores indicate better recovery.
Numerical rating scale score | changes of month 1, month 2 and month 3 after initial injection, and month 3 after final injection
  To assess pain relief of the knee joint. The numerical rating scale score ranges from 0-10, with a score of 0 indicating no pain and 10 indicating intense pain.

CONTACTS AND LOCATIONS:
Overall Officials: Quanyi Guo, Ph.D, Principal Investigator — Chinese PLA Hospital, China

IPD SHARING:
Plan to Share IPD: Undecided